CLINICAL TRIAL: NCT04991779
Title: A Multicenter Diagnostic Study on the Utility of AI-assisted Continue EEG Diagnosis of Neonatal Seizures
Brief Title: AI-assisted cEEG Diagnosis of Neonatal Seizures in Neonatal Intensive Care Unit
Status: Withdrawn | Type: Observational
Why Stopped: The other study was concluded as planned upon reaching its predetermined endpoint, which included the completion of data collection and achievement of the necessary sample size for statistical significance.
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Chengdu Women's and Children's Central Hospital (Other); Xiamen Children's Hospital (Other); Kunming Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHFudanU_NNICU16
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Neonatal Seizure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The neonates with suspected seizures or high risk of seizures: The neonates with suspected seizures or high risk of seizures are monitored by continuous electroencephalogram (cEEG) at least 12 hours since admission. The cEEG will be interpreted by AI-assisted cEEG diagnostic tool at the end of cEEG monitoring. At the same time, the same cEEG will be manually reported according the reference standard.
  Interventions: Diagnostic Test: AI-assisted cEEG detection tool

INTERVENTIONS:
Diagnostic Test: AI-assisted cEEG detection tool — This study is an observational study to evaluate the accuracy of AI-assisted cEEG diagnostic tool with routine care. All patients from the cohort accept cEEG monitoring and AI-assisted cEEG detection tool.
  The tool included a quantitive EEG neural signal processing pipeline to extract features from the original signal datasets, machine learning models based on gradient boosted model for prediction.
  The reference standard is the electrographic seizures interpreted by 3 clinicians who had attended the uniformly training program and were certified by the Chinese Anti-Epilepsy Association.

SUMMARY:
A diagnostic accuracy study on Artificial intelligence assisted continue EEG diagnostic tool is to carried out comparing with manually EEG interpretation as the golden standard for neonatal seizure.

DETAILED DESCRIPTION:
The occurrence of neonatal seizures may be the first, and perhaps the only, clinical sign of a central nervous system disorder in the newborn infant. The incidence of neonatal seizures is variable based on gestational age. The etiology of seizures may indicate the presence of a potentially treatable etiology and should prompt an immediate evaluation to determine the cause and to initiate etiology-specific therapy. Importantly, the earlier treatment of seizures positively affects the infant's long-term neurological development. However, even when continue electroencephalogram (cEEG) monitoring is available, the availability of on-site expertise to interpret cEEG signals is limited and in practice, the diagnosis is still based only on clinical signs. The previous study indicated that the reliable seizure detection was as little as 10% of seizure events. Therefore, an early automated seizure detection tool has been developed based on machine learning. The lack of an automated seizure detection tool has been validated in the external neonatal seizures cohort. The evidence on the utility of the automated seizure detection tool remains uncertain. This is a prospective, continuous double-blind designed diagnostic accuracy study. The study aims to validate the accuracy of the artificial intelligence (AI)-assisted cEEG diagnostic tool comparing the manually cEEG interpretation as the golden standard of neonatal seizure in neonatal intensive care units. Analysis of sensitivity and specificity is to evaluate the accuracy of AI-assisted cEEG diagnostic tool.

ELIGIBILITY:
Inclusion Criteria:

* Postnatal age < or = 28 days;
* cEEG monitoring at least 12hours monitoring;
* Suspected seizures;
* Risk of Intracranial hemorrhage;
* Abnormality of MRI or ultrasound before cEEG;
* Neonates diagnosed with encephalopathy or suspected of encephalopathy;
* Hypoxic-ischemic encephalopathy or suspected hypoxic-ischemic encephalopathy;
* Metabolic disturbances (Hypoglycemia, Hypocalcemia, Hypomagnesemia, Inborn errors of metabolism);
* Central nervous system (CNS) or systemic infections;
* Postsurgical neonatal within 3 days;
* Suspected genetic disease or Positive genetic diagnoses;

Exclusion Criteria:

* The neonates with head scalp defect, scalp hematoma, edema and other contraindications which are not suitable for cEEG monitoring during hospitalization.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with suspected seizures and high risk of seizures
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
The accuracy of AI-assisted cEEG diagnostic tool in evaluating the neonatal seizure | within 7 days since the end of cEEG monitoring during hospitalization
  The accuracy of includes sensitivity and specificity. The reference standard is the electrographic seizures interpreted by 3 clinicians who had attended the uniformly training program and were certified by the Chinese Anti-Epilepsy Association.
  Sensitivity is defined as: The proportion of neonates with seizures is successfully screened out by AI-assisted cEEG diagnostic tool.
  Specificity is defined as: The proportion of neonates without seizures who are not recognized as seizures by AI-assisted cEEG diagnostic tool.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, Ph.D, Study Chair — Children's Hospital of Fudan University
Locations (3):
- China (3):
  - Henan Children's Hospital, Zhengzhou, Henan
  - Children Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan

REFERENCES:
- [Result] Rennie JM, de Vries LS, Blennow M, Foran A, Shah DK, Livingstone V, van Huffelen AC, Mathieson SR, Pavlidis E, Weeke LC, Toet MC, Finder M, Pinnamaneni RM, Murray DM, Ryan AC, Marnane WP, Boylan GB. Characterisation of neonatal seizures and their treatment using continuous EEG monitoring: a multicentre experience. Arch Dis Child Fetal Neonatal Ed. 2019 Sep;104(5):F493-F501. doi: 10.1136/archdischild-2018-315624. Epub 2018 Nov 24. PMID 30472660
- [Result] Shellhaas RA, Chang T, Tsuchida T, Scher MS, Riviello JJ, Abend NS, Nguyen S, Wusthoff CJ, Clancy RR. The American Clinical Neurophysiology Society's Guideline on Continuous Electroencephalography Monitoring in Neonates. J Clin Neurophysiol. 2011 Dec;28(6):611-7. doi: 10.1097/WNP.0b013e31823e96d7. No abstract available. PMID 22146359
- [Result] Hoodbhoy Z, Masroor Jeelani S, Aziz A, Habib MI, Iqbal B, Akmal W, Siddiqui K, Hasan B, Leeflang M, Das JK. Machine Learning for Child and Adolescent Health: A Systematic Review. Pediatrics. 2021 Jan;147(1):e2020011833. doi: 10.1542/peds.2020-011833. Epub 2020 Dec 15. PMID 33323492